CLINICAL TRIAL: NCT03699774
Title: An Open-label, Fixed Sequence, Two-period Study to Evaluate the Effects of Repeated Doses of DS-8500a on the Pharmacokinetics of Rosuvastatin in Healthy Subjects.
Brief Title: Effect of Repeated Doses of DS-8500a on Pharmacokinetics of Rosuvastatin in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: DS8500-A-U105
Record Dates: First submitted 2018-10-05; First posted 2018-10-09 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2018-10

CONDITIONS: Drug Pharmacokinetics in Healthy Volunteers
MeSH Terms: interventions — firuglipel; Rosuvastatin Calcium

STUDY DESIGN:
Intervention Model Description: Fixed sequence
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- All Participants (Experimental): In treatment Period 1 (Day 1 through Day 4), on Day 1, participants receive a single dose of rosuvastatin 10 mg orally with food, and in Period 2 (Day 1 through Day 16), starting on Day 1, participants receive DS-8500a 75 mg orally qd with food for 16 days with concomitant administration of a single dose of rosuvastatin 10 mg qd on Day 14.
  In both the periods, rosuvastatin and DS-8500a are administered after an overnight fast of 8 hours and within 10 minutes after consuming a standardized breakfast of 500 calories.
  Interventions: Drug: DS-8500a; Drug: Rosuvastatin

INTERVENTIONS:
Drug: DS-8500a — DS-8500a is provided as three 25-mg tablets for oral administration
  Other Names: Experimental product
Drug: Rosuvastatin — Rosuvastatin is provided as a 10-mg tablet for oral administration
  Other Names: Crestor

SUMMARY:
The primary purpose of this study is to assess the effect of repeated doses of DS-8500a on the single dose pharmacokinetics (PK) of rosuvastatin.

The total length of time (from screening to follow-up) for each participant is approximately 7 weeks.

It is expected that repeated oral doses of DS-8500a will not have a significant effect on the pharmacokinetics of a single dose of rosuvastatin.

ELIGIBILITY:
Inclusion Criteria:

* Is healthy and of non-child-bearing potential
* Has a body mass index of 18-30 kg/m^2
* Has negative results for drugs of abuse, cotinine (smoking) and alcohol at screening
* Has signed informed consent and agreed to comply with all study requirements

Exclusion Criteria:

* Has history or current evidence of clinically significant cardiac, hepatic, renal, pulmonary, endocrine/metabolic, neurologic, infectious, gastrointestinal , hematologic, or oncologic disease as determined by screening history, physical examination, laboratory test results, or 12-lead ECG
* Has any other condition detailed in the protocol, or that in the opinion of the Investigator, precludes participation in the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-05-12 (Actual); Primary Completion 2015-07-06 (Actual); Study Completion 2015-07-06 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma drug concentration (Cmax) for single dose rosuvastatin | on Day 1 of Period 1 and Day 14 of Period 2
Time of maximum observed concentration (Tmax) for single dose rosuvastatin | on Day 1 of Period 1 and Day 14 of Period 2
Area under the plasma concentration time curve (AUC) from time 0 to the last quantifiable concentration (AUClast) for single dose rosuvastatin | on Day 1 of Period 1 and Day 14 of Period 2

SECONDARY OUTCOMES:
Cmax for DS-8500a and its metabolites | on Day 1 (for single dose) and Day 16 (for multiple dose) of Period 2
  Categories: DS-8500a, A209-3952, A210-2519, and A210-7951
Tmax for DS-8500a and its metabolites | on Day 1 (for single dose) and Day 16 (for multiple dose) of Period 2
  Categories: DS-8500a, A209-3952, A210-2519, and A210-7951
AUC from time 0 to 24 hours (AUC0-24) for DS-8500a and its metabolites | on Day 1 (for single dose) and Day 16 (for multiple dose) of Period 2
  Categories: DS-8500a, A209-3952, A210-2519, and A210-7951
Metabolite to parent (M:P) AUC0-24 ratios for DS-8500a and its metabolites | on Day 1 (for single dose) and Day 16 (for multiple dose) of Period 2
  Categories: A209-3952:DS-8500a, A210-2519:DS-8500a, and A210-7951:DS-8500a
Minimum observed analyte concentration that was just prior to the beginning of the dosing interval (Ctrough) | Days 2, 3, 5, 7, 10, 14, and 16 of Period 2
Cmax at steady state (Cmax,ss) | Day 16 of Period 2
AUC during the 24 hour dosing interval (AUCtau) | Day 16 of Period 2
Accumulation ratio (AccRatio) | Day 16 of Period 2
Tmax at steady state (Tmax,ss) | Day 16 of Period 2

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Leader, Study Director — Daiichi Sankyo
Locations (1):
- Worldwide Clinical Trials (WCT) Early Phase Services, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Maekawa Y, Furuie H, Kato M, Myobatake Y, Kamiyama E, Watanabe A, Shiosakai K, Taguchi T, Bass R, Zhou J, Dishy V, Warren V, Vashi V, Ishizuka H. Effect of DS-8500a, a Novel G Protein-Coupled Receptor 119 Agonist, on the Pharmacokinetics of Rosuvastatin and Atorvastatin in Healthy Subjects. Clin Drug Investig. 2019 Oct;39(10):967-978. doi: 10.1007/s40261-019-00825-1. PMID 31321631